CLINICAL TRIAL: NCT06214806
Title: Impact of a Food Purchasing Intervention on Consumption Patterns and Improved Dietary Outcomes in New Orleans - Food Is Medicine
Brief Title: Food Is Medicine: Makin' Healthy Groceries
Acronym: FIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Heart Association (Other); Rouses Market (Unknown); Instacart (Unknown); Duke Clinical Research Institute (Other); University Medical Center New Orleans - LCMC Health (Unknown); Louisiana Public Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00114628
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
Keywords: Food Insecurity; Food As Medicine; American Heart Association (AHA); New Orleans; Louisiana; PCORnet; Electronic Health Record (EHR); Cardiovascular Disease; Hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Food delivered via Instacart versus comparator arm of food purchased in-person at Rouses Market
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instacart (Experimental): Voucher for grocery purchase and delivery via Instacart
  Interventions: Behavioral: Grocery Vouchers
- Rouses Market (Active Comparator): Voucher for grocery purchase in-person at Rouses Market in New Orleans
  Interventions: Behavioral: Grocery Vouchers

INTERVENTIONS:
Behavioral: Grocery Vouchers — Participants will be given vouchers to buy groceries each month for five months.

SUMMARY:
This is a minimal risk study focusing on food purchasing and consumption in 100 subjects in the greater New Orleans area. There is evidence showing that individually-targeted vouchers effectively increase category-level food purchases in both less healthful and more healthful categories. This pilot study will investigate whether a voucher program using Instacart or a local, brick-and-mortar supermarket in New Orleans, LA lead to changes in food purchasing patterns, food consumption, food insecurity, and access to healthy food options for the participants, who are at risk of cardiovascular disease and/or cardiac complications. The study will also measure concordance between food purchasing and actual consumption.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 50 years of age
* Uncontrolled hypertension (defined as at least two clinically documented blood pressure readings of systolic BP >= 140 AND diastolic BP >=90 in the prior 6 months)
* Understands English

Exclusion Criteria:

* No internet access (at home, library, relative, or though phone plan)
* No adequate transportation (personal car, reliable ride, bus, and/or Uber/Lyft) in the New Orleans area

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Change in food consumption | Baseline, every month for 5 months
  Self-reported consumption of servings of fruits and vegetables combined, assessed through food frequency questionnaire

SECONDARY OUTCOMES:
Change in food purchasing | Every month, between months 1-5
  Imputed dollar amount spent on fruits and vegetables, derived from purchasing data
Use of voucher | Every month, between months 1-5
  Average dollar amount of voucher spent per month

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernandez, MD, MHS, Principal Investigator — Duke Clinical Research Institute; Thomas W Carton, PhD, MS, Study Director — Louisiana Public Health Institute (LPHI); Bridget Simon-Friedt, Study Chair — Louisiana Public Health Institute (LPHI)
Locations (2):
- United States (2):
  - University Medical Center New Orleans - LCMC Health, New Orleans, Louisiana
  - Louisiana Public Health Institute (LPHI), New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://storymaps.arcgis.com/stories/1a76c35080a8433487308f8526393b48